CLINICAL TRIAL: NCT05383508
Title: A Single-center, Randomized, Controlled, Open-label, Cross-over Study in Healthy Subjects to Investigate the Nicotine Pharmacokinetic Profiles of 2 Variants of P4M3 Gen 2.0, an Electronic Nicotine Delivery System, Compared to Cigarettes
Brief Title: Nicotine Pharmacokinetics Following Use of the P4M3 Gen 2.0 E-Cigarette Compared to Smoking Cigarettes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philip Morris Products S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: P4-PK-04-US
Record Dates: First submitted 2022-05-17; First posted 2022-05-20 (Actual); Results first posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Nicotine Vaping; Nicotine; Vaping
Keywords: Nicotine; Pharmacokinetics; Smoking; Cigarette; E-Cigarette
MeSH Terms: conditions — Vaping; Smoking | interventions — Fibronectins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Product Sequence 1 (Active Comparator): After at least 12 hours of abstinence from the use of any nicotine/tobacco containing products (referred to as nicotine wash-out), subjects will smoke a cigarette or use one of the e-liquid variants with P4M3 Gen 2.0 according to randomized product use sequence ad libitum for 6 minutes (± 30 seconds).
  CA35 on Day 1; Cig on Day 2; CM35 on Day 3
  Interventions: Other: CA35; Other: CM35; Other: Cig
- Product Sequence 2 (Active Comparator): After at least 12 hours of abstinence from the use of any nicotine/tobacco containing products (referred to as nicotine wash-out), subjects will smoke a cigarette or use one of the e-liquid variants with P4M3 Gen 2.0 according to randomized product use sequence ad libitum for 6 minutes (± 30 seconds).
  CA35 on Day 1; CM35 on Day 2; Cig on Day 3
  Interventions: Other: CA35; Other: CM35; Other: Cig
- Product Sequence 3 (Active Comparator): After at least 12 hours of abstinence from the use of any nicotine/tobacco containing products (referred to as nicotine wash-out), subjects will smoke a cigarette or use one of the e-liquid variants with P4M3 Gen 2.0 according to randomized product use sequence ad libitum for 6 minutes (± 30 seconds).
  Cig on Day 1; CA35 on Day 2; CM35 on Day 3
  Interventions: Other: CA35; Other: CM35; Other: Cig
- Product Sequence 4 (Active Comparator): After at least 12 hours of abstinence from the use of any nicotine/tobacco containing products (referred to as nicotine wash-out), subjects will smoke a cigarette or use one of the e-liquid variants with P4M3 Gen 2.0 according to randomized product use sequence ad libitum for 6 minutes (± 30 seconds).
  Cig on Day 1; CM35 on Day 2; CA35 on Day 3
  Interventions: Other: CA35; Other: CM35; Other: Cig
- Product Sequence 5 (Active Comparator): After at least 12 hours of abstinence from the use of any nicotine/tobacco containing products (referred to as nicotine wash-out), subjects will smoke a cigarette or use one of the e-liquid variants with P4M3 Gen 2.0 according to randomized product use sequence ad libitum for 6 minutes (± 30 seconds).
  CM35 on Day 1; Cig on Day 2; CA35 on Day 3
  Interventions: Other: CA35; Other: CM35; Other: Cig
- Product Sequence 6 (Active Comparator): After at least 12 hours of abstinence from the use of any nicotine/tobacco containing products (referred to as nicotine wash-out), subjects will smoke a cigarette or use one of the e-liquid variants with P4M3 Gen 2.0 according to randomized product use sequence ad libitum for 6 minutes (± 30 seconds).
  CM35 on Day 1; CA35 on Day 2; Cig on Day 3
  Interventions: Other: CA35; Other: CM35; Other: Cig

INTERVENTIONS:
Other: CA35 — Nicotine concentration: 3.5 % e-liquid flavor: Tobacco
  Other Names: P4M3 variant CA35
Other: CM35 — Nicotine concentration: 3.5 % e-liquid flavor: Menthol
  Other Names: P4M3 variant CM35
Other: Cig — Subjects' preferred brand of commercially available, regular or mentholated cigarettes

SUMMARY:
This is a single-center, randomized, controlled, open-label, cross-over study with healthy adult smokers. The study will investigate the nicotine pharmacokinetic (PK) profiles of two e-liquid variants used with the P4M3 Gen 2.0 e-cigarette, compared to smoking combustible cigarettes.

In addition, pharmacodynamic (PD) effects (subjective effects and related behavioral assessments), will be evaluated to provide further insights on product evaluation, craving, liking, puffing topography. The study will be conducted with three periods and six sequences in a cross-over design.

This study is exploratory and there is no pre-specified hypothesis to be tested.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate the nicotine pharmacokinetics (PK) profiles of two e-liquid variants used with the P4M3 Gen 2.0 e-cigarette versus cigarettes following a six minutes ad libitum use period. In addition, pharmacodynamic effects (PD), including subjective effects and related behavioral assessments, as well as human puffing topography (HPT) will be evaluated, to provide further insights on P4M3 Gen 2.0 product acceptance and product use. Safety will be assessed throughout the study.

The aim is to evaluate if P4M3 Gen 2.0 can provide an acceptable alternative to smoking cigarettes in terms of both, nicotine delivery and sensorial satisfaction for current adult smokers who would otherwise continue smoking cigarettes.

ELIGIBILITY:
Inclusion Criteria:

* Subject has signed the ICF and is able to understand the information provided in the ICF.
* Subject has smoked continuously for at least the last 3 years prior to the Screening visit.
* Subject has smoked ≥ 10 commercially available cigarettes per day for 4 weeks prior to Screening Visit and Admission.
* Subject does not plan to quit smoking cigarettes or using other nicotine or tobacco containing products in the next 3 months.
* Smoking, healthy subject as judged by the Investigator or designee based on available assessments from the Screening period.

Exclusion Criteria:

* As per the Investigator's judgment, the subject cannot participate in the study for any reason other than medical.
* Subject has donated or received whole blood or blood products within 30 days prior to Screening Visit.
* BMI < 18.5 kg/m2 or > 35.0 kg/m2.
* Subject has received medication within 14 days or within 5 half-lives of the drug prior to Admission (whichever is longer), which has an impact on CYP2A6 activity.
* Subject has a positive serology test for HIV 1/2, Hepatitis B or Hepatitis C.
* Subject has a history of alcohol abuse that could interfere with the subject's participation in study.
* Subject has a positive urine drug test.
* Subject has a positive alcohol breath test.
* Subject has participated in another clinical study within 30 days prior to the Screening Visit.
* Subject is pregnant (does not have negative pregnancy tests at Screening Visit and at Admission) or is breastfeeding.
* For women of childbearing potential only: subject does not agree to use an acceptable method of effective contraception.

Ages: 24 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2022-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Fein, MD, Principal Investigator — High Point Clinical Trials Center (HPCTC)
Locations (1):
- High Point Clinical Trials Center (HPCTC), High Point, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 36 subjects were enrolled in the study, which was conducted at a clinical trial facility managed by a contract research organization.
Pre-assignment Details: The 36 enrolled subjects were each randomized to one of six possible use sequences of product use.
Groups:
- Product Sequence 1: Subjects randomized to this product use sequence:
  CA35 on Day 1; Cig on Day 2; CM35 on Day 3
- Product Sequence 2: Subjects randomized to this product use sequence:
  CA35 on Day 1; CM35 on Day 2; Cig on Day 3
- Product Sequence 3: Subjects randomized to this product use sequence:
  Cig on Day 1; CA35 on Day 2; CM35 on Day 3
- Product Sequence 4: Subjects randomized to this product use sequence:
  Cig on Day 1; CM35 on Day 2; CA35 on Day 3
- Product Sequence 5: Subjects randomized to this product use sequence:
  CM35 on Day 1; Cig on Day 2; CA35 on Day 3
- Product Sequence 6: Subjects randomized to this product use sequence:
  CM35 on Day 1; CA35 on Day 2; Cig on Day 3
Period: Overall Study
Arm/Group | Product Sequence 1 | Product Sequence 2 | Product Sequence 3 | Product Sequence 4 | Product Sequence 5 | Product Sequence 6
Started | 6 | 6 | 6 | 6 | 6 | 6
Completed | 5 | 6 | 5 | 5 | 4 | 6
Not Completed | 1 | 0 | 1 | 1 | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Safety Population: Safety Population = All subjects who were exposed to the investigational product
Arm/Group | Safety Population
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (11.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 25
  White | 10
  Not Hispanic or Latino | 0
BMI [Mean (Standard Deviation); unit: kg/m²] | 29.783 (3.534)

OUTCOME MEASURES:

1. Primary Outcome: Background-corrected Maximum Plasma Concentration [Cmax]
Description: To measure Cmax from 6 minutes ad libitum use for two e-liquid variants used with the P4M3 Gen 2.0 e-cigarette and for subjects smoking cigarettes.
Time Frame: T0 = start of product use. From day 1 to day 3, blood was drawn 5 minutes prior to T0 (day 1 only), and then 1, 2, 4, 6, 8, 10, 12, 15, 30 minutes, 1, 2, 4, 10 and 24 hours after T0. (Note that sample taken 24 hours after T0 on day 1 and day 2 only.)
Population: The analysis population was a subset of the Safety Population and consisted of all randomized subjects, without major protocol deviations, for whom at least one nicotine PK parameter could be derived.
Measure: Geometric Mean (95% Confidence Interval); unit: (ng/mL)
Groups:
- CA35: P4M3 Gen 2.0 Classic Auburn 3.5% nicotine
- CM35: P4M3 Gen 2.0 Classic Menthol 3.5% nicotine
- Cigarettes: Subject's own cigarettes
Arm/Group | CA35 | CM35 | Cigarettes
Number analyzed (Participants) | 22 | 23 | 23
(ng/mL) | 2.934 [1.695 to 5.080] | 3.365 [1.919 to 5.900] | 17.49 [12.29 to 24.89]
Statistical Analysis 1: Comparison: CA35 vs Cigarettes; The objective of this study was to determine the Cmax ratio of P4M3 variants:Cigarettes along with the corresponding 95% confidence intervals; Test type: Other; Mixed Models Analysis — 95% confidence intervals are provided for this analysis; The model included terms for sequence, period, and product exposure as fixed effects and subject as a categorical random effect; Geometric LS Mean Ratio (%) = 17.05, 95% CI 2-sided [10.69 to 27.19] — Analysis was performed on log transformed data with Kenward Roger degrees of freedom approximation. Ratio and related 95% CI were derived by exponentiating the estimates obtained on the log scale
Statistical Analysis 2: Comparison: CM35 vs Cigarettes; [analysis description as in outcome 1, analysis 1]; Test type: Other; Mixed Models Analysis — 95% confidence intervals are provided for this analysis; [statistical method as in outcome 1, analysis 1]; Geometric LS Mean Ratio (%) = 19.47, 95% CI 2-sided [11.89 to 31.87] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Background-corrected Time to the Maximum Concentration [Tmax]
Description: To measure Tmax from 6 minutes ad libitum use for two e-liquid variants used with the P4M3 Gen 2.0 e-cigarette and for subjects smoking cigarettes.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | CA35 | CM35 | Cigarettes
Number analyzed (Participants) | 22 | 23 | 23
minutes | 109.3 [-33.28 to 251.8] | 37.79 [-15.62 to 91.21] | 7.826 [6.926 to 8.726]
Statistical Analysis 1: Comparison: CA35 vs Cigarettes; The objective of this study was to determine the Tmax difference of P4M3 variants:Cigarettes along with the corresponding 95% confidence intervals; Test type: Other; Wilcoxon signed rank test — 95% confidence intervals are provided for this analysis; Median Difference (Net) = 3.000, 95% CI 2-sided [0.00 to 11.00] — Hodges-Lehmann estimator of location shift and Moses 95% CI
Statistical Analysis 2: Comparison: CM35 vs Cigarettes; [analysis description as in outcome 2, analysis 1]; Test type: Other; Wilcoxon signed rank test — 95% confidence intervals are provided for this analysis; Mean Difference (Net) = 2.000, 95% CI 2-sided [0.00 to 4.00] — Hodges-Lehmann estimator of location shift and Moses 95% CI

3. Primary Outcome: Area Under the Background-corrected Concentration-time Curve From Start of Product Use to Time of Last Quantifiable Concentration and Extrapolated to Infinity.
Description: To measure the area under the background-corrected concentration-time curve (AUC) from start of product use from 6 minutes ad libitum use for two e-liquid variants used with the P4M3 Gen 2.0 e-cigarette and for subjects smoking cigarettes.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: min*ng/mL
Arm/Group | CA35 | CM35 | Cigarettes
Number analyzed (Participants) | 14 | 14 | 19
min*ng/mL | 891.1 [515.6 to 1540] | 655.6 [317.0 to 1356] | 2484 [1880 to 3283]
Statistical Analysis 1: Comparison: CA35 vs Cigarettes; The objective of this study was to determine the AUC0-infinity ratio of P4M3 variants:Cigarettes along with the corresponding 95% confidence intervals; Test type: Other; Mixed Models Analysis — 95% confidence intervals are provided for this analysis; [statistical method as in outcome 1, analysis 1]; Geometric LS Mean Ratio (%) = 28.29, 95% CI 2-sided [16.00 to 50.04] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: CM35 vs Cigarettes; [analysis description as in outcome 3, analysis 1]; Test type: Other; Mixed Models Analysis — 95% confidence intervals are provided for this analysis; [statistical method as in outcome 1, analysis 1]; Geometric LS Mean Ratio (%) = 26.16, 95% CI 2-sided [12.74 to 53.69] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Maximum Ratio of Background-corrected Concentration Over Time
Description: To measure the maximum ratio of background-corrected concentration over time, from T0 (excluded) to Tmax (included)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: (ng/mL)/min
Arm/Group | CA35 | CM35 | Cigarettes
Number analyzed (Participants) | 22 | 23 | 23
(ng/mL)/min | 0.3547 [0.1618 to 0.7777] | 0.5150 [0.2760 to 0.9610] | 3.239 [2.277 to 4.608]
Statistical Analysis 1: Comparison: CA35 vs Cigarettes; The objective of this study was to determine the maximum ratio of background-corrected concentration over time of P4M3 variants:Cigarettes along with the corresponding 95% confidence intervals; Test type: Other; Mixed Models Analysis — 95% confidence intervals are provided for this analysis; [statistical method as in outcome 1, analysis 1]; Geometric LS Mean Ratio (%) = 10.84, 95% CI 2-sided [5.57 to 21.10] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: CM35 vs Cigarettes; [analysis description as in outcome 4, analysis 1]; Test type: Other; Mixed Models Analysis — 95% confidence intervals are provided for this analysis; [statistical method as in outcome 1, analysis 1]; Geometric LS Mean Ratio (%) = 16.83, 95% CI 2-sided [9.93 to 28.53] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the signature of the ICF by each subject until the end of the safety follow-up period, a total duration for each subject of up to 34 days.
Groups:
- Safety Population (CA35 Test); Safety Population (CA35); Safety Population (CM35); Cigarettes: The safety population was a subset of the screened population and consisted of all subjects who gave informed consent, had at least one exposure to P4M3 Gen 2.0, including the product test at Admission (Day -1), and had at least one safety assessment.
Arm/Group | Safety Population (CA35 Test) | Safety Population (CA35) | Safety Population (CM35) | Cigarettes
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/32 | 0/33 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/32 | 0/33 | 0/34
Other Adverse Events (participants affected / at risk) | 0/35 | 0/32 | 0/33 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
We confirm we have the contractual provisions in place which specify that in no event will the study site be allowed to disclose to any third party (or publicly release) any information obtained through the study without the CRO's prior written consent which in turn cannot provide such consent without Sponsor's approval unless such publication is made to satisfy regulatory requirements.

The Intellectual Property rights and research results from the present study belong to the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2021-10-14): https://cdn.clinicaltrials.gov/large-docs/08/NCT05383508/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/08/NCT05383508/SAP_001.pdf